CLINICAL TRIAL: NCT02301663
Title: DEVELOPMENT OF A NOVEL STRESS TESTING PROTOCOL TO DEFINE THE RELATIONSHIP BETWEEN CORONARY MICROVASCULAR DYSFUNCTION AND DIASTOLOGY IN WOMEN WITH ANGINA BUT NO EVIDENCE OF OBSTRUCTIVE CORONARY ARTERY DISEASE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Diastolic stress testing
Record Dates: First submitted 2014-11-22; First posted 2014-11-26 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Microvascular Coronary Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Women w/microvascular disease (Experimental): 10 women with microvascular disease
  Interventions: Other: Handgrip; Other: Altitude simulation; Other: Leg exercise
- Normal controls (Experimental): 10 age-matched women with no evidence of microvascular disease
  Interventions: Other: Handgrip; Other: Altitude simulation; Other: Leg exercise
- calibration (Experimental): 10 healthy individuals who will help to synchronize our imaging and stress testing maneuvers.
  Interventions: Other: Handgrip; Other: Altitude simulation; Other: Leg exercise

INTERVENTIONS:
Other: Handgrip — Subjects will be asked to squeeze and handgrip dynamometer to increase cardiac metabolic demand
Other: Altitude simulation — Subjects will breathe a lower concentration of oxygen to simulate the effects of altitude.
Other: Leg exercise — Subjects will perform leg exercise to increase metabolic demand.

SUMMARY:
Microvascular coronary dysfunction (MCD) (abnormities in small blood vessels/arteries in heart) with symptoms of persistent chest pain, primarily impacts women. There are an estimated 2-3 million women in the US with MCD and about 100,000 new cases annually. Recent data from our research group suggests that coronary microvascular disease impairs the way the heart relaxes. This pilot study will attempt to exacerbate this phenotype in an effort to better understand the pathophysiology of the disease. The investigators will recruit 30 volunteers total (10 healthy calibration subjects, 10 women with microvascular disease, and 10 age-match women for the group with microvascular disease). Subjects will undergo a series of "stress" maneuvers in conjunction with advanced cardiac magnetic resonance imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understanding and willing to undergo study procedures
2. Male or Female greater than or equal to 18 years of age
3. Understanding and willing to sign consent form.

Exclusion Criteria:

1. History of cardiovascular, pulmonary, or neurological disease
2. Hypertension (sitting blood pressure >140/90 mmHg, with measurements recorded on at least 2 occasions)
3. Diabetes
4. Unable to give informed consent;
5. Contra-indication to CMRI testing, including claustrophobia and metallic implants
6. Adherence or retention issues;
7. Women who are pregnant.
8. Allergy to animal dander.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2030-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Diastolic function by MRI | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Michael Nelson, PhD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes